CLINICAL TRIAL: NCT05766033
Title: Bracket Failure Rate With a Novel Etchant Paste. A Randomized Clinical Trial
Brief Title: Bracket Failure With a Novel Etchant Paste. A Randomized Clinical Trial
Acronym: failurerate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hussein Qays Aswad, hqaswad, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Bracket failure rate
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Orthodontic Appliance Complication

STUDY DESIGN:
Intervention Model Description: This is a multi-center, single-operator, split-mouth randomized controlled trial with a 1:1 allocation ratio.
Who Masked: Investigator
Masking Description: Allocation concealment is achieved with sequentially numbered, opaque sealed envelopes containing the side allocation of the etchant, prepared before the trial. An independent person is responsible for opening the next envelope in sequence and implementing the randomization process. Blinding of the operator at bracket bonding is not possible because of the nature of the intervention. Blinding of the patient is not considered relevant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel etchent paste (Experimental)
  Interventions: Other: Enamel conditioning with a novel etchant paste
- Phosphoric acid 37% (Active Comparator)
  Interventions: Other: Enamel conditioning with a novel etchant paste

INTERVENTIONS:
Other: Enamel conditioning with a novel etchant paste — The maxillary and mandibular incisors, canines, and premolars for each patient will be conditioned using the Novel etchent paste on one side (experimental), while the other side (control) conditioned with a phosphoric acid gel 37% . Both systems use identical brackets and adhesive system (differ only with regard to the etching system).
  Other Names: Etching for enamel for bracket bonding

SUMMARY:
To investigate metallic brackets failure rate bonded post enamel conditioning with a novel CaP etchant paste in comparison with those bonded following conventional enamel etching with PA gel over a period of 6 months.

DETAILED DESCRIPTION:
Acid etching of tooth surfaces to promote the bonding of orthodontic attachments to the enamel has been a routine procedure in orthodontic treatment since the 1960s. Various types of orthodontic etchants and etching techniques have been introduced in the past five decades. Michael G Buonocore in revolutionized dentistry with his historical paper: "A simple method of increasing the adhesion of acrylic filling materials to enamel surfaces" depicting the advantage of etching and bonding of acrylic to enamel. It forever changed the practice of dentistry. Buonocore and Silverstone led the profession in acid etching and bonding of resin to etched enamel surfaces. These developments allowed orthodontists to bond brackets reliably and apply forces to move teeth without banding every tooth or having brackets deboned. Buonocore reported that 85% phosphoric acid etchant significantly increased the adhesion of acrylic resin to enamel. Since then, a variety of etchants have been used with different concentrations and etching times. These include hydrofluoric acid, citric acid, hydrochloric acid, maleic acid, nitric acid, and phosphoric acid in a variety of concentrations. Suggested etching times can vary from 15 to 60 seconds. The tooth enamel surface is known for its low-energy and hydrophobic properties, with its outermost layer being rich in fluoride. Enamel etching with phosphoric acid (PA) removes the fluoride-rich layer, dissolves enamel mineral, creates micro- pores, and renders a high-energy and hydrophilic enamel surface to permit wetting by an adhesive; yet at the expense of increased surface porosity, susceptibility to staining, caries, more remnant adhesive and enamel loss. Fixation of brackets to teeth involves joining of two different solid substrates or adherents through an intervening adhesive layer. Bracket bases are currently provided with mesh designs that ensure robust mechanical interlocking between the bracket and adhesive, whilst research is ongoing to improve enamel conditioning strategies that can attain clinically successful bond strengths yet maintain an unblemished enamel surface. Alternative methods to conventional enamel etching with phosphoric acid have been sought aiming at decreasing the bond strength to reduce the incidence of enamel damage. The use of glass ionomer cements for orthodontic bonding decreased the occurrence of enamel damage, yet at the expense of clinically unacceptable bond strengths. On the other hand, the use of laser etching and self- etch primers resulted in bracket shear bond strengths comparable to the conventional etch-and-rinse approach, but could not eliminate enamel damage. In 2019, Ibrahim et al developed a new bioactive orthodontic etchant paste made of calcium-phosphate (CaP), which could alleviate subsurface enamel demineralization in comparison with the traditional phosphoric acid etchant and the pre-clinical viability assessment using in vitro studies showed exemplary advantages. The new low-pH CaP paste etchant application is a clinically viable bracket bonding method with steps similar to PA application that yielded adequate bond strength with the advantages of minimal adhesive remnants and no enamel chipping or cracking on deboning of the bracket.

ELIGIBILITY:
Inclusion Criteria.

* Full permanent dentition including incisors, canines, premolars, and ﬁrst molars.
* Teeth with sound, non-carious buccal enamel and no pretreatment with chemical agents such as hydrogen peroxide.
* No previous orthodontic treatment with ﬁxed appliances.

Exclusion Criteria:

* Were unable to give informed consent) Had craniofacial anomalies.
* Required orthognathic surgery as part of their treatment.
* Had congenital enamel defects

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Bracket failure rate | 6 months
  Patients with repeated bond failures caused by habits or trauma would be excluded from further analysis.only counting the number of brackets that broken .

SECONDARY OUTCOMES:
Adhesive remenant index | 6 months
  Assessment of the amount of remnant adhesive left post bracket failure (for both methods).This index system was developed on the basis of a pilot study of 20 extracted teeth and the criteria were as follows: score 0 = no adhesive left on the tooth; score 1 = less than half of the adhesive left on the tooth; score 2 = more than half of the adhesive left on the tooth; and score 3 = all adhesive left on the tooth with a distinct impression of the bracket mesh.

CONTACTS AND LOCATIONS:
Locations (1):
- Hussain Qays Aswad, Baghdad, Alrusafaa, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
till now there is no plan to share it when i found it i will updated it.

REFERENCES:
- [Background] Ibrahim AI, Al-Hasani NR, Thompson VP, Deb S. Resistance of bonded premolars to four artificial ageing models post enamel conditioning with a novel calcium-phosphate paste. J Clin Exp Dent. 2020 Apr 1;12(4):e317-e326. doi: 10.4317/jced.56764. eCollection 2020 Apr. PMID 32382380